CLINICAL TRIAL: NCT00296179
Title: Comparison of Zolpidem Tartrate Extended-Release vs. Placebo in Treatment of Insomnia Associated With Newly Diagnosed Major Depressive Disorder(MDD) or Untreated MDD Relapse, When Used Concomitantly With Escitalopram
Brief Title: Ambien CR For Treatment Of Insomnia Associated With Depression When Used Concomitantly With Lexapro
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PM_L_0166
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2008-07-28 (Estimated); Status verified 2008-07

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

INTERVENTIONS:
Drug: zolpidem tartrate

SUMMARY:
To demonstrate overall improvement of insomnia in subjects treated with zolpidem tartrate extended-release (Ambien CR) and escitalopram (Lexapro) vs. subjects treated with placebo and escitalopram at 2 months.

ELIGIBILITY:
MAJOR INCLUSION CRITERIA:

1. Must experience sleep disturbances at least 3 nights/week, based on historical data
2. Must meet the diagnostic requirements for Major Depressive Disorder
3. Must have QIDS-SR16 score between 6 and 15
4. Must be either newly diagnosed or show symptoms of relapse/recurrence of depression while not on medication
5. Age 21-64, inclusive
6. Women must use a medically acceptable form of contraception (steroidal contraceptive, double-barrier, or intra-uterine device) during the entire study period, or: be surgically sterilized, post-menopausal, agree to use double-barrier contraception throughout the study period, or must have a negative urine pregnancy test prior to randomization.
7. Subject must be stabilized on all ongoing long-term medication therapy for at least 28 days prior to screening visit.

MAJOR EXCLUSION CRITERIA:

1. Severity of depressive episode had been rated as "severe" or "severe with psychotic features."
2. History of a suicide attempt or suicidal ideation.
3. History of mania, manic episode or bipolar disease.
4. Currently using a benzodiazepine or SSRI or more than 2 days of use within the 28 days preceding randomization.
5. Use of prescription and non-prescription sedative drugs given for the purpose of sleep induction or to relieve jet lag
6. Any abnormal pre-study laboratory values that require clinical intervention
7. Prior failure to respond to escitalopram therapy for depression
8. Current depressive episode requiring inpatient hospitalization.
9. Shift work or requirement for a regular change in sleep schedule by at least six hours within the previous 28 days.
10. History of drug addiction, alcoholism, or drug abuse.
11. A positive urine drug screen for medication that would interfere with the assessment of the study medication.
12. Known allergy to zolpidem, escitalopram or any of their excipients
13. History of sleep apnea
14. History of myasthenia gravis
15. The presence of any untreated or uncompensated clinically significant renal, endocrine, gastrointestinal, hepatic, respiratory, cardiovascular, other neurologic, hematologic, oncologic, immunologic, cerebrovascular disease or malignancy.
16. Pregnant or breastfeeding
17. Subject is participating in another clinical trial, or has completed another clinical trial within 28 days prior to screening.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 372
Dates: Start 2006-02; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Efficacy: Patient-reported TST

SECONDARY OUTCOMES:
Difference in relapse rates in patients receiving placebo and patients receiving zolpidem MR during 4 month follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, Study Director — Sanofi

REFERENCES:
- [Derived] Fava M, Asnis GM, Shrivastava RK, Lydiard B, Bastani B, Sheehan DV, Roth T. Improved insomnia symptoms and sleep-related next-day functioning in patients with comorbid major depressive disorder and insomnia following concomitant zolpidem extended-release 12.5 mg and escitalopram treatment: a randomized controlled trial. J Clin Psychiatry. 2011 Jul;72(7):914-28. doi: 10.4088/JCP.09m05571gry. Epub 2010 Dec 28. PMID 21208597